CLINICAL TRIAL: NCT07362914
Title: The Role of Corticosteroids in Hand & Foot & Skin Reactions Reduction to Doxorubicin Liposomes
Brief Title: Corticosteroids for Doxorubicin Liposome-Induced Hand-Foot-Skin Reactions
Acronym: CHORD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2412310-10
Record Dates: First submitted 2025-05-11; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A(NEO-DXMS GROUP) (Experimental): no dexamethasone
  Interventions: Drug: Doxorubicin hydrochloride liposome injection; Drug: Cyclophosphamide
- Arm B( MED-DEX GROUP ) (Experimental): dexamethasone 12mg d1, PO/IV
  Interventions: Drug: Dexamethasone (12mg d1); Drug: Doxorubicin hydrochloride liposome injection; Drug: Cyclophosphamide
- Arm C(HIGH-DEX GROUP ) (Experimental): dexamethasone 12mg QD, d1-5, PO/IV
  Interventions: Drug: Dexamethasone (2mg QD, d1-5,); Drug: Doxorubicin hydrochloride liposome injection; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Dexamethasone (12mg d1) — dexamethasone 12mg d1, PO/IV;
  Arms: Arm B( MED-DEX GROUP )
Drug: Dexamethasone (2mg QD, d1-5,) — dexamethasone 12mg QD, d1-5, PO/IV.
  Arms: Arm C(HIGH-DEX GROUP )
Drug: Doxorubicin hydrochloride liposome injection — Liposomal doxorubicin at a dose of 35 mg/m², given via intravenous (IV) infusion every 2 weeks (q2w) or every 3 weeks (q3w).
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m² administered by intravenous infusion every 2 weeks (q2w) or every 3 weeks (q3w).

SUMMARY:
Investigating the Association Between Corticosteroid Use and Improvement in Doxorubicin Liposome-Induced Cutaneous Toxicity: Exploring the Feasibility and Mechanisms of Corticosteroids in Mitigating Liposomal Doxorubicin-Related Dermatologic Adverse Effects.

DETAILED DESCRIPTION:
Background

Liposomal doxorubicin exhibits distinct toxicity profiles compared to free-form doxorubicin in clinical practice. Cutaneous toxicity represents the primary dose-limiting adverse effect of liposomal doxorubicin, with incidence and severity demonstrating a dose-dependent relationship . Current management strategies-including dose reduction or extended treatment intervals-yield limited efficacy, often leading to treatment discontinuation due to intolerable symptoms, thereby compromising clinical utility.

Mechanistic Insights

Our preliminary research identified neutrophils as key mediators in liposomal skin accumulation:

Complement receptor 3 (CR3) recognizes iC3b deposited on liposomes via complement activation.

Neutrophils phagocytose liposomes and extravasate into cutaneous tissues, driving drug accumulation.

Intervention with complement inhibitors significantly reduced liposomal doxorubicin deposition in murine skin by:

Blocking complement activation Decreasing iC3b opsonization Inhibiting neutrophil-mediated uptake.

Clinical Evidence

A retrospective study at our center demonstrated that corticosteroid pretreatment alleviated liposomal doxorubicin-induced hand-foot syndrome (HFS) in a dose-dependent manner :

High-dose corticosteroids limited Grade 1 HFS to <10% of patients16. Findings support complement inhibition as a viable strategy for mitigating cutaneous toxicity7.

Study Objectives

This prospective study aims to:

Correlate corticosteroid use with HFS severity reduction in liposomal doxorubicin therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years (inclusive), regardless of gender.
2. Diagnosis & Treatment Plan: Histopathologically confirmed early-stage or advanced breast cancer patients eligible for AC regimen (liposomal doxorubicin + cyclophosphamide) chemotherapy per clinical guidelines.
3. ECOG Performance Status: Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
4. Anticipated survival ≥3 months.
5. Organ Function Requirements:

   Hematologic: Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L ,Platelet count ≥75 × 10⁹/L Hemoglobin ≥90 g/L

   Hepatic:

   Non-liver metastasis: Total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN Liver metastasis: TBIL ≤1.5 × ULN ,ALT and AST ≤5 × ULN

   Renal:

   Serum creatinine (Cr) ≤1.5 × ULN or creatinine clearance (Ccr) ≥50 mL/min

   Coagulation:

   International normalized ratio (INR) or prothrombin time (PT) ≤1.5 × ULN Activated partial thromboplastin time (APTT) ≤1.5 × ULN
6. Contraception:

   Female patients: Must use effective contraception (e.g., intrauterine device [IUD], oral contraceptives, or condoms) during the study and for 6 months after study completion. A negative serum pregnancy test within 7 days prior to enrollment is required, and patients must be non-lactating.

   Male patients: Must agree to use contraception during the study and for 6 months after study completion.
7. Informed Consent: Patients must voluntarily participate, provide signed informed consent, and comply with protocol-specified procedures (blood tests, follow-ups, etc.).

Exclusion Criteria:

1. Received chemotherapy, radiotherapy, biologics, targeted therapy, immunotherapy, or other antitumor treatments within 4 weeks before the first study dose (or within 5 half-lives, whichever is shorter). Exceptions: The washout period may be adjusted per investigator judgment (e.g., shortened to 2 weeks for endocrine therapy to avoid prolonged patient waiting).
2. Previous treatment with liposomal doxorubicin or similar formulations.
3. Allergy History: Known hypersensitivity to liposomal products or doxorubicin.
4. Cardiovascular Diseases:

   Severe arrhythmias/conduction abnormalities (e.g., clinically significant ventricular arrhythmias, second- or third-degree AV block).

   History of myocardial infarction, coronary artery bypass grafting (CABG), or heart failure (NYHA Class ≥II).

   LVEF ≤50%or prolonged QTcF (>450 ms in males; >470 ms in females).
5. Active Infections: Grade ≥2 （NCI CTCAE v5.0）
6. Immunosuppression:

   Active autoimmune diseases, immunodeficiency (e.g., HIV-positive), or congenital/acquired immune disorders.

   History of organ transplantation or chronic corticosteroid use.
7. HBsAg-positive with HBV-DNA ≥500 IU/mL. Exception: If HBV-DNA <500 IU/mL and chronic hepatitis is deemed stable/inactive by the investigator, enrollment is permitted.
8. Other Infections: Positive for HCV antibody or syphilis-specific antibody.
9. Neurological/Psychiatric Disorders: History of epilepsy, dementia, or other uncontrolled conditions.
10. CNS Metastases: Symptomatic brain or leptomeningeal metastases, or uncontrolled CNS lesions. Exception: Asymptomatic brain metastases or lesions stable for ≥28 days without steroids/antitumor therapy are allowed.
11. Any other condition that, per investigator assessment, may compromise patient safety or study compliance.
12. Pregnant or breastfeeding women.
13. Patients deemed ineligible for the study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with hand-foot syndrome (HFS) as assessed by CTCAE v5.0 in the high-dose dexamethasone group | 17 months
  Compared to both the no-dexamethasone group and the standard-dose dexamethasone group, the high-dose dexamethasone group demonstrated reduced incidence of hand-foot syndrome (HFS)

SECONDARY OUTCOMES:
ncidence of Treatment-Emergent Adverse Events | 17 months
  Standardized terminology for dermatologic adverse events, typically graded per CTCAE (Common Terminology Criteria for Adverse Events) v5.0 criteria
Disease-free survival (DFS) | 17 months
  Defined as the time from randomization (or treatment initiation in single-arm trials) to disease recurrence or death from any cause.
Progression-free survival (PFS) | 17 months
  The duration from treatment initiation to tumor progression (per RECIST 1.1 ) or death.
Overall survival (OS) | 17 months
  Time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No